CLINICAL TRIAL: NCT02807441
Title: Association Between Perioperative Bleeding and Aspirin Use in Spine Surgery: A Randomized, Controlled Trial
Brief Title: Perioperative Bleeding and Aspirin Use in Spine Surgery
Acronym: ASA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Heather Fuhrman, medical student, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UHCMC-Ortho
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Hemorrhage; Thrombosis
Keywords: Bleeding; Aspirin; Spine; Surgery
MeSH Terms: conditions — Hemorrhage; Thrombosis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No aspirin (No Intervention): Patients will not be given any Acetylsalicylic acid in the perioperative period.
- Low-dose aspirin (Experimental): Patients will be given low-dose Acetylsalicylic acid (81 mg) in the perioperative period.
  Interventions: Drug: Acetylsalicylic acid
- High-dose aspirin (Experimental): Patients will be given high-dose Acetylsalicylic acid (325 mg) in the perioperative period.
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Acetylsalicylic acid — Patients will receive different doses of aspirin perioperatively to assess bleeding association.
  Other Names: aspirin
  Arms: High-dose aspirin; Low-dose aspirin

SUMMARY:
The investigators would like to further the current understanding of aspirin and its effects on perioperative bleeding by conducting a randomized controlled trial of spinal surgery patients receiving varying doses of aspirin or no aspirin perioperatively. The investigators hypothesize that there will be no significant difference in perioperative blood loss between the different groups.

DETAILED DESCRIPTION:
Selected patients will be given either no aspirin, low-dose aspirin (81 mg), or high-dose aspirin (325 mg) in the perioperative period. These dosages are based on the Pharmacist's letter/Prescriber's letter which provides aspirin dosing recommendations for varying cardiovascular indications. Allocation of dosing will be based on computerized randomization in order to achieve approximately 100 patients in each group. Patient records will then be assessed for demographic characteristics, comorbidities, symptoms, functional outcome scores (Sf-12), operative time, intraoperative estimated blood loss, postoperative blood loss in drainage tubes (when applicable), cumulative blood loss, transfusion of blood products, hemoglobin level, preoperative International Normalized Ratio (INR), preoperative platelet count, hospital length of stay, and morbidity and mortality including development of NSTEMI, atrial fibrillation, surgical site infection, pulmonary embolism, and hospital 30-day readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old, who are not taking aspirin at the time of operation as part of a current cardiovascular treatment plan, who will undergo spinal surgery from 2016-2019 in the practice of Dr. Eubanks.

Exclusion Criteria:

* Any patient under the age of 18 and/or is already taking anticoagulant therapy for an established cardiovascular disease at the time of surgery as part of a cardiovascular therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Hemorrhage: Amount of blood loss | Intraoperative
  Amount of blood loss from the operation will be recorded
Hemorrhage: Amount of blood loss | 48 hours Postoperative
  Blood loss from drainage tube when applicable

SECONDARY OUTCOMES:
Blood Transfusion: Amount of blood products transfused | Intraoperative
  Amount of blood products transfused when applicable

CONTACTS AND LOCATIONS:
Overall Officials: Jason Eubanks, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be collected on a computer database containing unique identifiers, without names, social security numbers, medical record numbers, or other information that could be used to identify individuals. University Hospitals Research Electronic Data Capture will be used as a means of secure data storage. At no time will this data spreadsheet be printed or otherwise distributed, and no Protected Health Information will be transferred to investigators at other sites of this multi-center study.

REFERENCES:
- [Background] Hall R, Mazer CD. Antiplatelet drugs: a review of their pharmacology and management in the perioperative period. Anesth Analg. 2011 Feb;112(2):292-318. doi: 10.1213/ANE.0b013e318203f38d. Epub 2011 Jan 6. PMID 21212258
- [Background] Cuellar JM, Petrizzo A, Vaswani R, Goldstein JA, Bendo JA. Does aspirin administration increase perioperative morbidity in patients with cardiac stents undergoing spinal surgery? Spine (Phila Pa 1976). 2015 May 1;40(9):629-35. doi: 10.1097/BRS.0000000000000695. PMID 26030214
- [Background] Gerstein NS, Schulman PM, Gerstein WH, Petersen TR, Tawil I. Should more patients continue aspirin therapy perioperatively?: clinical impact of aspirin withdrawal syndrome. Ann Surg. 2012 May;255(5):811-9. doi: 10.1097/SLA.0b013e318250504e. PMID 22470078
- [Background] Soleman J, Baumgarten P, Perrig WN, Fandino J, Fathi AR. Non-instrumented extradural lumbar spine surgery under low-dose acetylsalicylic acid: a comparative risk analysis study. Eur Spine J. 2016 Mar;25(3):732-9. doi: 10.1007/s00586-015-3864-7. Epub 2015 Mar 11. PMID 25757534
- [Background] Gerstein NS, Carey MC, Cigarroa JE, Schulman PM. Perioperative aspirin management after POISE-2: some answers, but questions remain. Anesth Analg. 2015 Mar;120(3):570-575. doi: 10.1213/ANE.0000000000000589. PMID 25695574
- [Background] Manchikanti L, Abdi S, Atluri S, Benyamin RM, Boswell MV, Buenaventura RM, Bryce DA, Burks PA, Caraway DL, Calodney AK, Cash KA, Christo PJ, Cohen SP, Colson J, Conn A, Cordner H, Coubarous S, Datta S, Deer TR, Diwan S, Falco FJ, Fellows B, Geffert S, Grider JS, Gupta S, Hameed H, Hameed M, Hansen H, Helm S 2nd, Janata JW, Justiz R, Kaye AD, Lee M, Manchikanti KN, McManus CD, Onyewu O, Parr AT, Patel VB, Racz GB, Sehgal N, Sharma ML, Simopoulos TT, Singh V, Smith HS, Snook LT, Swicegood JR, Vallejo R, Ward SP, Wargo BW, Zhu J, Hirsch JA. An update of comprehensive evidence-based guidelines for interventional techniques in chronic spinal pain. Part II: guidance and recommendations. Pain Physician. 2013 Apr;16(2 Suppl):S49-283. PMID 23615883
- [Background] Park HJ, Kwon KY, Woo JH. Comparison of blood loss according to use of aspirin in lumbar fusion patients. Eur Spine J. 2014 Aug;23(8):1777-82. doi: 10.1007/s00586-014-3294-y. Epub 2014 Apr 17. PMID 24740280
- [Background] Kang SB, Cho KJ, Moon KH, Jung JH, Jung SJ. Does low-dose aspirin increase blood loss after spinal fusion surgery? Spine J. 2011 Apr;11(4):303-7. doi: 10.1016/j.spinee.2011.02.006. PMID 21474081
- [Background] Wong SS, Irwin MG. Peri-operative cardiac protection for non-cardiac surgery. Anaesthesia. 2016 Jan;71 Suppl 1:29-39. doi: 10.1111/anae.13305. PMID 26620144